CLINICAL TRIAL: NCT06537323
Title: Comparative Analysis of Educational Interventions and Anesthetic Techniques for Enhanced Spinal Anesthesia Quality in Fractured Neck of Femur: Femoral Nerve Block, Periarticular Nerve Group (PENG) Block, and Preoperative IV Fentanyl
Brief Title: Femoral Nerve Block, Periarticular Nerve Group (PENG) Block, and Preoperative IV Fentanyl
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Zaher Zaki Zaher, Lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Aswu 918/5/24
Record Dates: First submitted 2024-07-25; First posted 2024-08-05 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Femoral nerve block with0.25% bupivacaine (Other): Femoral nerve block with0.25% bupivacaine guided by ultrasound.
  Interventions: Drug: Femoral nerve block with0.25% bupivacaine guided by ultrasound.
- PENG block with0.25% bupivacaine (Other): PENG block with0.25% bupivacaine guided by ultrasound
  Interventions: Drug: PENG block with0.25% bupivacaine guided by ultrasound.
- Preoperative IV fentanyl (Other): Preoperative IV fentanyl 100microgram
  Interventions: Drug: Preoperative IV fentanyl 100microgram

INTERVENTIONS:
Drug: Femoral nerve block with0.25% bupivacaine guided by ultrasound. — Femoral nerve block with0.25% bupivacaine guided by ultrasound.
  Arms: Femoral nerve block with0.25% bupivacaine
Drug: PENG block with0.25% bupivacaine guided by ultrasound. — PENG block with0.25% bupivacaine guided by ultrasound.
  Arms: PENG block with0.25% bupivacaine
Drug: Preoperative IV fentanyl 100microgram — Preoperative IV fentanyl 100microgram
  Arms: Preoperative IV fentanyl

SUMMARY:
The pericapsular nerve group block is a regional anesthetic technique described in 2018, developed primarily in total hip arthroplasties for postoperative analgesia with motor sparing benefits. The block is thought to provide more complete analgesia to the hip by depositing local anesthetic within the myofascial plane of the psoas muscle and superior pubic ramus. The indications for total hip arthroplasties often include degenerative hip disease and traumatic hip fractures. These indications for surgery are relatively common in the elderly population and are associated with significant morbidity and mortality.

DETAILED DESCRIPTION:
The pericapsular nerve block is a regional anesthetic technique described in 2018, developed primarily in total hip arthroplasties for postoperative analgesia with motor sparing benefits. The block is thought to provide more complete analgesia to the hip by depositing local anesthetic within the myofascial plane of the psoas muscle and superior pubic ramus.The indications for total hip arthroplasties often include degenerative hip disease and traumatic hip fractures. These indications for surgery are relatively common in the elderly population and are associated with significant morbidity and mortality.Operative intervention, such as total hip arthroplasties has also been associated with significant pain. Historically, the most commonly performed peripheral nerve blocks include lumbar plexus block, a femoral nerve block, or a fascia iliaca compartment block to manage post-operative analgesia. With the understanding that additional articular branches these blocks will provide incomplete analgesia to the hip and may also predispose the patient to fall due to weakness of the quadriceps muscles.Therefore the ideal block technique should provide complete analgesia of the hip joint and without muscle weakness. The ultrasound-guided pericapsular nerve block block allows for coverage of the hip joint, targeting the proximal articular branches that innervate the joint capsule. This proximal approach via ultrasound guidance can confer several advantages over a femoral nerve block by providing more complete analgesia to the hip joint. Additionally, the motor function of the involved extremity should be spared. The pericapsular nerve block block can be used alone as a primary analgesic or in conjunction with other forms of anesthesia during surgery or in the perioperative period. For lateral surgical incisions, a supplemental lateral femoral cutaneous nerve block provides additional coverage.The femoral nerve is among the largest branches of the lumbar plexus. The femoral nerve arises from the ventral rami of the Lumeber 2, Lumber 3, and Lumber 4 spinal nerves, and enters the femoral triangle inferior to the inguinal ligament. The femoral nerve is the most lateral of the structures within the triangle, which also contains the femoral artery and femoral vein at its medial end. The femoral nerve splits into anterior and posterior divisions that originate near the level of the circumflex artery. The anterior division gives rise to the medial femoral cutaneous nerve and innervates the sartorius muscle. The posterior division gives rise to the saphenous nerve and provides innervation to quadriceps femoris muscle. In addition to motor innervation, the femoral nerve provides sensation to the anterior thigh and knee and the medial lower extremity below the knee. The saphenous nerve is a femoral nerve branch that is directly responsible for sensation to the medial lower leg and foot. The saphenous nerve can be blocked separately at the level of the adductor canal, and several more distal sites. The adductor canal is a musculoaponeurotic tunnel found in the mid-thigh and extends from the femoral triangle to the adductor magnus.Due to the anatomical connection, the femoral nerve within the femoral triage may potentially be affected by proximal or high-volume adductor canal blocks.

ELIGIBILITY:
Inclusion Criteria:

* The included patient should be between 55 to 69 years

Exclusion Criteria:

* known allergies to local anesthetics

Ages: 55 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
EOSA score (Ease of Spinal Anesthesia) Score | before procedure, 24 hours and 30 days
  Ease of Spinal Anesthesia (EOSA) Score The Ease of Spinal Anesthesia (EOSA) score is a structured tool used to evaluate the technical ease and patient cooperation during spinal anesthesia administration. It incorporates multiple factors that influence the success and efficiency of the procedure.
  Components of the EOSA Score:
  The score assesses the following five key factors:
  Patient positioning time - The time required to achieve an optimal position for spinal anesthesia.
  Patient cooperation - The level of patient compliance and ability to maintain the required position.
  Technical difficulty - The ease of needle insertion, including the number of attempts required.
  Need for additional assistance - Whether repositioning, sedation, or extra staff intervention was required.
  Anesthesiologist's overall ease rating - The subjective assessment of how smoothly the procedure was performed.
  Each factor is assigned a score, with higher EOSA scores indicating greater ease of spinal anesthesia a

SECONDARY OUTCOMES:
time to the first request for analgesia, nalbuphine consumption within the first 24 hours, postoperative pain scores, intraoperative hemodynamic stability, duration of the spinal block, patient satisfaction, the incidence of complications, | before procedure, 24 hours and 30 days,VAS at 1, 6, 12, and 24 hours postoperatively.-Hemodynamic parameters, including mean arterial blood pressure (MAP) and heart rate (HR), were recorded at baseline, and subsequently at 30, 60, 90, and 120 minutes, as
  Hemodynamic parameters, including mean arterial blood pressure (MAP) and heart rate (HR), were recorded at baseline, and subsequently at 30, 60, 90, and 120 minutes, as well as at the end of surgery.
  Pain was evaluated using VAS at 1, 6, 12, and 24 hours postoperatively. The total amount of nalbuphine used during the first 24 hours. If the VAS score exceeded 4, 0.1 mg/kg nalbuphine was administered. The time to first rescue analgesia was measured from the end of surgery to the initial request for additional pain relief.
  Complications, including hypotension, nausea, vomiting, respiratory depression, pruritus, urinary retention, motor weakness, local anesthetic systemic toxicity, and block-related side effects, were meticulously documented. Hypotension, a reduction in baseline means arterial pressure by 20% or an absolute value below 65 mmHg, was managed with 10 mg of ephedrine. Postoperative nausea and vomiting (PONV) were treated with intravenous ondansetron at a dose of 0.1 mg/kg.
BMI | At base line
  Weight in Kg /(height in meter *height in meter)
  =kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Zaher, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No